CLINICAL TRIAL: NCT05514366
Title: Influence of Inspiratory Pause on Ventilatory Efficiency and Tidal Volume Distribution in Patients Undergoing Robotic Prostate Surgery and Ventilated With an Individualized Open Lung Approach. A Prospective Paired Study.
Brief Title: Influence of Inspiratory Pause on Ventilatory Efficiency in Robotic Surgery. A Prospective Paired Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIP2022.FISEVI
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Mechanical Ventilation; Positive End-Expiratory Pressure; Anesthesia
Keywords: Intermittent Positive-Pressure Ventilation; Positive End-Expiratory Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- End inspiratory pause under tOLA (Experimental): Application of four different end inspiratory pauses (EIP) corresponding to 10, 20, 30 and 40% of inspiratory time.
  Phase 1) before the application of pneumoperitoneum and forced trendelenburg. Phase 2) during the application of pneumoperitoneum and forced trendelenburg. During both phases, all patients will be ventilated under a tOLA strategy (see Study Description section).
  Interventions: Procedure: Modifying EIP under a tOLA before pneumoperitoneum; Procedure: Modifying EIP under a tOLA with pneumoperitoneum; Procedure: Atelectasis test

INTERVENTIONS:
Procedure: Modifying EIP under a tOLA before pneumoperitoneum — Phase 1:
  Moment (M) 1) Standard PPV and an initial EIP of 10%
  M 2) ARM with titration of optimal PEEP (PEEPop) on a decremental PEEP trial, followed by a new ARM and setting a tailored open-lung PEEP (tOL-PEEP), that 2 cm H2O higher than PEEPop
  M 3) Incremental modification of the EIP in steps of 10% (from 10 to 40%)
Procedure: Modifying EIP under a tOLA with pneumoperitoneum — Phase 2:
  M 4) The investigators will apply the EIP that guarantees the lowest Pdriv
  M 5) After applying pneumoperitoneum and trendelenburg
  M 6) Atelectasis test (see below)
  M 7) M 7a) In case of atelectasis test = negative: the investigators will modify the EIP in incremental or decremental steps of 10% M 7b) In case of atelectasis test=positive: ARM
  M 8) In those cases recruited (M 7b), modify the EIP (as in M 7a)
  Once the EIP that guarantees the best ventilation conditions has been stablished based on the lowest Pdriv (and higher Crs), the investigators will maintain these conditions until the end of surgery, with periodic evaluation of the pulmonary collapse by means of the atelectasis test (see below) performed every 40 minutes or regardless of time if an oxygen saturation by pulse oximetry (SpO2) < 97% is detected.
Procedure: Atelectasis test — It is performed during mechanical ventilation, due to suspicion of alveolar collapse. Alveolar collapse will be suspected on observation of a reduction in Crs > 10% over post-recruitment values. In these cases the atelectasis test will be performed, consisting of a reduction in FiO2 to 0.21, maintaining this FiO2 for 5 minutes. If lung collapse is >10%, a fall in SpO2 below 97% will be expected (positive atelectasis test), in which case, an ARM and a PEEPop titration test will be performed.

SUMMARY:
The investigators aim to determine if the modification of the end inspiratory pause (EIP) during mechanical ventilation adds benefit when applied to patients undergoing robotic surgery and who are ventilated under an individualized open lung approach (iOLA) strategy. The EIP is an adjustable parameter of volume controlled ventilation modes usually set as a percentage of the total inspiratory time. It represents the phase comprised between the moment in which the volume programmed in the ventilator has already been administered (which marks the end of the inspiratory flow), and the opening of the expiratory valve (which marks the beginning of expiration).

The investigators will study whether modifications of the EIP produce variations in the "quantity" of the lung that participates in gas exchange (respiratory volume). To do so, the investigators will sequentially apply different EIP to participants (paired study). The investigators´ hypothesis is that increasing the EIP up to a level, may diminish the lung volume that does not participate in breathing (the physiological dead space- VDphys), thereby increasing the respiratory volume. To note: the VDphys includes the "conduction" volume, that represented by trachea, bronchi, et cetera, which is in charge of driving the "air" towards the respiratory zones, and the alveolar dead space (those zones of the respiratory volume that due to different reasons do not directly participate in gas exchange: alveoli ventilated but not perfused, areas of overdistension, etc. The investigators will measure dead volumes by mean of specific non-invasive monitoring (volumetric capnography) coupled to the anesthesia workstation, and the mechanics of lung and the distribution of the gas within it by means of electric impedance tomography, a non-invasive technique showing continuous images of patient's lung. The estimation of the respiratory volume will help the investigators to more precisely adjust the amount of oxygen and anesthetic gases that must be administered in function of patients´ gases consumption, a calculated parameter that is function of the respiratory volume and that will also be tested during the study. The investigators will also accurately measure patient oxygenation by means of arterial blood samples extracted from a radial artery catheter. Apart from sequential modifications in the EIP, the ventilation strategy applied to patients will be that used in the investigators´ usual practice (described below).

DETAILED DESCRIPTION:
Introduction

Mechanical ventilation (MV) during general anesthesia entails some adverse effects that cannot be completely avoided. In recent years, pulmonary protective ventilation (PPV) strategies, based on the use of a low tidal volume (TV) with the intention of reducing the biological trauma associated to MV, are gaining prominence in surgical and intensive care patients. A tailored open-lung approach (tOLA) has recently emerged as one of these PPV strategies. It combines the use of alveolar recruitment manoeuvers (ARM), aiming to "open" collapsed areas of the lung, with the application of individualised positive end expiratory pressure (PEEP) with the objective of avoiding the re-collapse of those areas during expiration. The rationale supporting OLA strategies assumes that achieving more homogeneous alveolar ventilation by preventing atelectasis, while avoiding alveolar overdistension, leads to a more efficient gas distribution and exchange. This allows less traumatic ventilation and reduces the inflammatory response. The use of a tOLA has shown promising results in terms of improving oxygenation and reducing the risk of severe postoperative pulmonary complications.

Along with the above, prolonging the end inspiratory pause (EIP), while maintaining an adequate expiratory time, has shown benefits in terms of improving effective alveolar ventilation and enhancing gas exchange. The investigators recently demonstrated the effects of increasing the EIP when ventilating patients with a tOLA strategy. In that work, the investigators examined the effects of two EIP (10 and 30% of the inspiratory time) on the respiratory mechanics of patients undergoing major surgery. The investigators studied the effect of EIP on driving pressure (Pdriv), plateau pressure (Pplat), compliance of the respiratory system (Crs) and PEEP. The investigators also evaluated the dynamic distribution of TV during the ventilatory cycle using electrical impedance tomography (EIT) and studied the effect of EIP on gas exchange by means of arterial gasometry. In that study, the benefits of a longer EIP were seen with both standard PPV (TV of 7 mL of predicted body weight (PBW) and a PEEP of 5 cmH2O), and with a tOLA. The tOLA strategy was associated with a significant increase in PEEP, Pplat, arterial pressure of oxygen (PaO2), and Crs, with a significant decrease in Pdriv and arterial pressure of carbon dioxide (PaCO2), and with a more homogeneous gas distribution compared to standard PPV. On the other hand, the use of a longer EIP showed a significantly lower PEEP, Pdriv and mean airway pressure (Pmean) together with a higher Crs among patients ventilated under a tOLA strategy. However, it was not an objective of the addressed work to study the effects of the EIP modification on ventilatory efficiency, measured as the relation between VDphys and TV (VDphys/TV), something that the investigators will address in this work.

The investigators hypothesize that increasing the EIP in the context of a tOLA may improve alveolar ventilation by reducing the VDphys/TV ratio; in other words, by reducing the dead volume. To test this hypothesis, the investigators will study patients submitted to abdominal robotic surgery. The investigators´ intention is to verify if the potential benefits associated with the combined use of a tOLA and a longer EIP are observed in this type of surgery, where the gas insufflated into the abdomen together with the surgical position (forced trendelenburg) are known to jeopardize ventilation conditions.

Methods

Prospective, paired study with consecutive recruitment of participants to be carried out in a tertiary care teaching hospital (Hospital Universitario Virgen del Rocío). Approval for this study will be sought from the local ethics committee. The recruitment will be made on investigators availability.

Study protocol. Following standard monitoring on arrival to the operating room, participants will be slightly sedated with intravenous midazolam 1-2 mg and remifentanil infusion 0.03-0.05 µg/kg/min The left radial artery will be catheterized under local anesthesia. For EIT monitoring, the PulmoVista 500 system (Dräger, Lübeck, Germany) will be used. Four regions of interest (ROI) will be defined as quadrants one through four, corresponding to top left and right (one, two) and bottom left and right (three, four). Global and regional impedance waveforms will be displayed continuously. The distribution of ventilation by ROI will be expressed as the regional proportion of gas distribution relative to total lung ventilation. Baseline data will be recorded during full consciousness with 0.21 fraction of inspired oxygen (FiO2). The investigators will then pre-oxygenate the participants through a face mask for 5 min in spontaneous ventilation with FIO2 of 0.8 and a fresh gas flow of 6 L/min. Anesthesia induction will performed with propofol (1-1.5 mg/kg PBW) and rocuronium 0.8 mg/kg PBW, proceeding with tracheal intubation. Patients will be ventilated through a Primus anesthesia workstation (Drager, Telford, PA, USA) using a TV of 7 mL/kg PBW. The ventilation mode used will be volume control, which will include an inspiration: expiration ratio of 1:2 and a respiratory rate of 12-15 breaths/min to maintain CO2 at the end of expiration between 35 and 40 mmHg and an initial PEEP of 5 cmH2O. A 10% EIP will be scheduled for all participants. A fresh gas flow of 0.5 to 1 L/min with an FIO2 of 0.5 will be used throughout the procedure. Anesthesia will be maintained with remifentanil 0.03 to 0.05 µg/kg/min and sevoflurane, with a minimum alveolar concentration of 0.6 to 0.8, which will be adjusted to the patient's age to ensure a Bispectral Index (BIS Quatro; Covidien Ilc , Mansfield, MA, USA) between 40-60. Rocuronium will be administered to ensure deep neuromuscular blockade during the study, which will be monitored by train of four neuromuscular relaxation (TOF-watch®, Organon Ltd., Swords, Co. Dublin, Ireland). All ventilation parameters will remain stable throughout the study except PEEP, which will be titrated according to the principles of tOLA, and EIP, which will be modified according to the study protocol (see Arms and Interventions section). Airway pressure (Paw), esophageal pressure (Pes) and gas flow will be measured with a Fluxmed® monitor (MBMED, Buenos Aires, Argentina). The data will be downloaded to a laptop after proper calibration of the flow and pressure sensors. The computer, through the FluxView software (MBMED, Buenos Aires, Argentina), will automatically calculate the following parameters:alveolar, airway and physiological dead volumes (VDalv, VDaw and VDphys, respectively) and its values related to the TV. Airway resistance (Raw = Ppeak-Pplat/inspiratory flow) will also be recorded, where Ppeak is peak pressure. A Pes measurement catheter (MBMED, Buenos Aires, Argentina) will be placed in the mid-esophageal position. Its position will be checked using the occlusion method described for patients with mechanical ventilation35. An acceptable catheter position will be found when the ΔPes/ΔPaw ratio is close to 1. Transpulmonary pressure (PTP) will be calculated as the difference between Paw and Pes. Transpulmonary driving pressure (PTPdriv) will be calculated as end-inspiratory transpulmonary pressure (PTPei) minus end-expiratory transpulmonary pressure (PTPee). Lung stress will be defined as PTPei. The elastance of the respiratory system (Ers= Pplat-PEEP/ TV) will be divided into its lung (El = Plei- Plee / TV) and chest wall (Ecw = Pesei- Pesee/TV) components. The anesthesia workstation will be used for continuous monitoring of Ppeak, Pplat, PEEP, Crs, FiO2 and CO2 at the end of expiration. An ABL90 FLEX PLUS device (Radiometer Medical, Copenhagen, Denmark) will be used for gas analysis.

Study sequence (detailed in the Arms and Interventions section):

Phase 1) The investigators will evaluate the impact of modifying the EIP (10 to 40%) in patients ventilated under an tOLA strategy before the instauration of surgical pneumoperitoneum.

Phase 2) The investigators will evaluate the impact of robotic conditions (pneumoperitoneum + forced trendelenburg) while applying different EIPs (10 to 40%).

Statistical analysis will be performed by the principal investigator. For data analysis, the statistical software IBM SPSS Statistics for Windows, version 24 (IBM Corp., Armonk, NY, USA) will be used. The investigators will perform an exploratory analysis of the data, using the mean ± standard deviation or the median with interquartile range for quantitative variables, and using percentages for the analysis of qualitative variables. The normality of data distribution will be checked with the Kolmogorov-Smirnov test or with the Shapiro-Wilk test for variables with less than 50 records. The Student's t test for paired samples will be used to study the behavior of the quantitative variables at different times (intragroup comparisons).

Calculation of the sample size was carried out by the main investigator, using version 4.2 of the EPIDAT statistical program (General Directorate of Innovation and Public Health Management of the Health Council of the Galician Government). The sample size was calculated based on the data from the previous work of the researchers, in which the investigators studied the influence of EIP on respiratory mechanics and the distribution of TV in surgical patients ventilated under an tOLA strategy (REF). The sample size was estimated assuming the differences in Crs when going from an EIP of 10% to 30% (paired sample). The investigators determined an average difference of 17 mL/cm H2O between both interventions. The sample size was calculated to obtain a power of 80% to detect differences in the contrast of the null hypothesis h₀: μ₁ = μ₂ using a two-sided Student's t-test for two related samples, considering a significance level of 5% and assuming the respective standard deviation in each group. Taking into account an expected percentage of dropouts of 20%, the sample size has been estimated at 17 pairs of experimental units under study (17 participants with paired treatment in the sample).

Amendment - Clarification of Sample Size Estimation

The original sample size calculation, as registered, was based on expected changes in Crs with different EIP settings, using data from a previous study by the investigators. This calculation was performed a priori using EPIDAT 4.2, and it remains valid for the Crs outcome.

However, during study execution, it became clear that the primary outcome of interest-VDphys-was insufficiently supported by published data, making the a priori estimation less precise for this variable. To address this, and after enrolling the first six subjects, the study team performed an unplanned, data-driven sample size re-estimation using G*Power 3.1.9.7, based on the observed mean difference in VDphys between EIP settings.

This re-estimation did not result in a change to the target sample size, which remained at 17 participants. We acknowledge that this procedure was not pre-specified in the original protocol and represents a methodological limitation. The deviation has been transparently reported and discussed in the revised manuscript.

The study continues to adhere to its original objectives, design, and statistical endpoints, and no other changes have been made to the methodology or outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years) scheduled for robotic prostatic surgery at the investigators´ institution
* Written informed consent

Exclusion Criteria:

* Participation in another interventional study
* Participants unable to understand the information contained in the informed consent
* American Society of Anesthesiologists (ASA) classification grade = IV
* Patient in dialysis
* Chronic obstructive pulmonary disease (COPD) grade Global Initiative for Chronic Obstructive Lung Disease(GOLD) > 2
* Functional vital capacity < 60% or > 120% of the predicted
* Body mass index (BMI) > 35 kg/m2
* Relation PaO2/FiO2 <200 mmHg in the baseline sample
* Presence of mechanical ventilation in the 72 hours prior to enrollment
* New York Heart Association (NYHA) functional class ≥ 3
* Clinically suspected heart failure
* Diagnosis or suspicion of intracranial hypertension
* Presence of pneumothorax or giant bullae on preoperative imaging tests
* Use of Continuous Positive Airway Pressure (CPAP).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in physiological dead space volume (VDphys) | Through the study completion: assessed in moments 1, 2, 3, 5, 7a and 8
  VDphys is that percentage of the tidal volume not participating of gas exchange

SECONDARY OUTCOMES:
Changes in intra-tidal gas distribution | Through the study completion: assessed in moments 1, 2, 3, 5, 7a and 8
  The distribution of the tidal gas within the lung during mechanical ventilation will be evaluated by means of EIT. It will be expressed as percentage of tidal gas distribution per region of interest (ROI).
Changes in arterial partial pressure of oxygen | Through the study completion: assessed in moments 1, 3, 7b and 8
  The investigators will measure patient oxygenation by means of arterial blood samples extracted from a radial artery catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel de la Matta, MD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
All the IPD collected, suitably anonymized, will be available to other researchers upon request by email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After finishing data analysis
Access Criteria: Upon other researchers request, through mail contact with the principal researcher

REFERENCES:
- [Background] Ladha K, Vidal Melo MF, McLean DJ, Wanderer JP, Grabitz SD, Kurth T, Eikermann M. Intraoperative protective mechanical ventilation and risk of postoperative respiratory complications: hospital based registry study. BMJ. 2015 Jul 14;351:h3646. doi: 10.1136/bmj.h3646. PMID 26174419
- [Background] Hemmes SN, Serpa Neto A, Schultz MJ. Intraoperative ventilatory strategies to prevent postoperative pulmonary complications: a meta-analysis. Curr Opin Anaesthesiol. 2013 Apr;26(2):126-33. doi: 10.1097/ACO.0b013e32835e1242. PMID 23385321
- [Background] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Moine P, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network investigators. Incidence of mortality and morbidity related to postoperative lung injury in patients who have undergone abdominal or thoracic surgery: a systematic review and meta-analysis. Lancet Respir Med. 2014 Dec;2(12):1007-15. doi: 10.1016/S2213-2600(14)70228-0. Epub 2014 Nov 13. PMID 25466352
- [Background] Futier E, Constantin JM, Jaber S. Protective lung ventilation in operating room: a systematic review. Minerva Anestesiol. 2014 Jun;80(6):726-35. Epub 2013 Nov 13. PMID 24226493
- [Background] Guay J, Ochroch EA. Intraoperative use of low volume ventilation to decrease postoperative mortality, mechanical ventilation, lengths of stay and lung injury in patients without acute lung injury. Cochrane Database Syst Rev. 2015 Dec 7;(12):CD011151. doi: 10.1002/14651858.CD011151.pub2. PMID 26641378
- [Background] Wolthuis EK, Choi G, Dessing MC, Bresser P, Lutter R, Dzoljic M, van der Poll T, Vroom MB, Hollmann M, Schultz MJ. Mechanical ventilation with lower tidal volumes and positive end-expiratory pressure prevents pulmonary inflammation in patients without preexisting lung injury. Anesthesiology. 2008 Jan;108(1):46-54. doi: 10.1097/01.anes.0000296068.80921.10. PMID 18156881
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Petrucci N, De Feo C. Lung protective ventilation strategy for the acute respiratory distress syndrome. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD003844. doi: 10.1002/14651858.CD003844.pub4. PMID 23450544
- [Background] Ferrando C, Suarez-Sipmann F, Tusman G, Leon I, Romero E, Gracia E, Mugarra A, Arocas B, Pozo N, Soro M, Belda FJ. Open lung approach versus standard protective strategies: Effects on driving pressure and ventilatory efficiency during anesthesia - A pilot, randomized controlled trial. PLoS One. 2017 May 11;12(5):e0177399. doi: 10.1371/journal.pone.0177399. eCollection 2017. PMID 28493943
- [Background] Ferrando C, Soro M, Canet J, Unzueta MC, Suarez F, Librero J, Peiro S, Llombart A, Delgado C, Leon I, Rovira L, Ramasco F, Granell M, Aldecoa C, Diaz O, Balust J, Garutti I, de la Matta M, Pensado A, Gonzalez R, Duran ME, Gallego L, Del Valle SG, Redondo FJ, Diaz P, Pestana D, Rodriguez A, Aguirre J, Garcia JM, Garcia J, Espinosa E, Charco P, Navarro J, Rodriguez C, Tusman G, Belda FJ; iPROVE investigators (Appendices 1 and 2). Rationale and study design for an individualized perioperative open lung ventilatory strategy (iPROVE): study protocol for a randomized controlled trial. Trials. 2015 Apr 27;16:193. doi: 10.1186/s13063-015-0694-1. PMID 25927183
- [Background] Ferrando C, Aldecoa C, Unzueta C, Belda FJ, Librero J, Tusman G, Suarez-Sipmann F, Peiro S, Pozo N, Brunelli A, Garutti I, Gallego C, Rodriguez A, Garcia JI, Diaz-Cambronero O, Balust J, Redondo FJ, de la Matta M, Gallego-Ligorit L, Hernandez J, Martinez P, Perez A, Leal S, Alday E, Monedero P, Gonzalez R, Mazzirani G, Aguilar G, Lopez-Baamonde M, Felipe M, Mugarra A, Torrente J, Valencia L, Varon V, Sanchez S, Rodriguez B, Martin A, India I, Azparren G, Molina R, Villar J, Soro M; iPROVE-O2 Network. Effects of oxygen on post-surgical infections during an individualised perioperative open-lung ventilatory strategy: a randomised controlled trial. Br J Anaesth. 2020 Jan;124(1):110-120. doi: 10.1016/j.bja.2019.10.009. Epub 2019 Nov 22. PMID 31767144
- [Background] Ferrando C, Mugarra A, Gutierrez A, Carbonell JA, Garcia M, Soro M, Tusman G, Belda FJ. Setting individualized positive end-expiratory pressure level with a positive end-expiratory pressure decrement trial after a recruitment maneuver improves oxygenation and lung mechanics during one-lung ventilation. Anesth Analg. 2014 Mar;118(3):657-65. doi: 10.1213/ANE.0000000000000105. PMID 24557111
- [Background] Ferrando C, Soro M, Unzueta C, Suarez-Sipmann F, Canet J, Librero J, Pozo N, Peiro S, Llombart A, Leon I, India I, Aldecoa C, Diaz-Cambronero O, Pestana D, Redondo FJ, Garutti I, Balust J, Garcia JI, Ibanez M, Granell M, Rodriguez A, Gallego L, de la Matta M, Gonzalez R, Brunelli A, Garcia J, Rovira L, Barrios F, Torres V, Hernandez S, Gracia E, Gine M, Garcia M, Garcia N, Miguel L, Sanchez S, Pineiro P, Pujol R, Garcia-Del-Valle S, Valdivia J, Hernandez MJ, Padron O, Colas A, Puig J, Azparren G, Tusman G, Villar J, Belda J; Individualized PeRioperative Open-lung VEntilation (iPROVE) Network. Individualised perioperative open-lung approach versus standard protective ventilation in abdominal surgery (iPROVE): a randomised controlled trial. Lancet Respir Med. 2018 Mar;6(3):193-203. doi: 10.1016/S2213-2600(18)30024-9. Epub 2018 Jan 19. PMID 29371130
- [Background] Maisch S, Reissmann H, Fuellekrug B, Weismann D, Rutkowski T, Tusman G, Bohm SH. Compliance and dead space fraction indicate an optimal level of positive end-expiratory pressure after recruitment in anesthetized patients. Anesth Analg. 2008 Jan;106(1):175-81, table of contents. doi: 10.1213/01.ane.0000287684.74505.49. PMID 18165575
- [Background] Williams EC, Motta-Ribeiro GC, Vidal Melo MF. Driving Pressure and Transpulmonary Pressure: How Do We Guide Safe Mechanical Ventilation? Anesthesiology. 2019 Jul;131(1):155-163. doi: 10.1097/ALN.0000000000002731. PMID 31094753
- [Background] Aboab J, Niklason L, Uttman L, Kouatchet A, Brochard L, Jonson B. CO2 elimination at varying inspiratory pause in acute lung injury. Clin Physiol Funct Imaging. 2007 Jan;27(1):2-6. doi: 10.1111/j.1475-097X.2007.00699.x. PMID 17204030
- [Background] Aboab J, Niklason L, Uttman L, Brochard L, Jonson B. Dead space and CO(2) elimination related to pattern of inspiratory gas delivery in ARDS patients. Crit Care. 2012 Dec 12;16(2):R39. doi: 10.1186/cc11232. PMID 22390777
- [Background] Aguirre-Bermeo H, Moran I, Bottiroli M, Italiano S, Parrilla FJ, Plazolles E, Roche-Campo F, Mancebo J. End-inspiratory pause prolongation in acute respiratory distress syndrome patients: effects on gas exchange and mechanics. Ann Intensive Care. 2016 Dec;6(1):81. doi: 10.1186/s13613-016-0183-z. Epub 2016 Aug 24. PMID 27558174
- [Background] Devaquet J, Jonson B, Niklason L, Si Larbi AG, Uttman L, Aboab J, Brochard L. Effects of inspiratory pause on CO2 elimination and arterial PCO2 in acute lung injury. J Appl Physiol (1985). 2008 Dec;105(6):1944-9. doi: 10.1152/japplphysiol.90682.2008. Epub 2008 Sep 18. PMID 18801962
- [Background] Uttman L, Jonson B. A prolonged postinspiratory pause enhances CO2 elimination by reducing airway dead space. Clin Physiol Funct Imaging. 2003 Sep;23(5):252-6. doi: 10.1046/j.1475-097x.2003.00498.x. PMID 12950321
- [Background] Sturesson LW, Malmkvist G, Allvin S, Collryd M, Bodelsson M, Jonson B. An appropriate inspiratory flow pattern can enhance CO2 exchange, facilitating protective ventilation of healthy lungs. Br J Anaesth. 2016 Aug;117(2):243-9. doi: 10.1093/bja/aew194. PMID 27440637
- [Background] Lopez-Herrera D, De La Matta M. Influence of the end inspiratory pause on respiratory mechanics and tidal gas distribution of surgical patients ventilated under a tailored open lung approach strategy: A randomised, crossover trial. Anaesth Crit Care Pain Med. 2022 Apr;41(2):101038. doi: 10.1016/j.accpm.2022.101038. Epub 2022 Feb 17. PMID 35183806
- [Background] Tusman G, Acosta CM, Ochoa M, Bohm SH, Gogniat E, Martinez Arca J, Scandurra A, Madorno M, Ferrando C, Suarez Sipmann F. Multimodal non-invasive monitoring to apply an open lung approach strategy in morbidly obese patients during bariatric surgery. J Clin Monit Comput. 2020 Oct;34(5):1015-1024. doi: 10.1007/s10877-019-00405-w. Epub 2019 Oct 25. PMID 31654282